CLINICAL TRIAL: NCT06669143
Title: The Efficacy and Safety of Zanubutinib-based for Post-remission Maintenance in Patients With Diffuse Large B-cell Lymphoma Who Are Intolerant to Intense First-line Chemotherapy
Brief Title: Zanubrutinib-based Maintenance Therapy of Newly Diagnosed DLBCL With Initial Remission
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zanubrutinib-based maintenance
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; zanubrutinib; maintenance
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib and Lenalidomide (Experimental)
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg bid, po, day 1-21, a maximum of 2 years.
Drug: Lenalidomide — 25 mg qd, po, day 1-10, a maximum of 2 years.

SUMMARY:
This single-arm, prospective clinical study will evaluate the efficacy and safety of Zanubrutinib-based maintenance therapy for post-remission in newly diagnosed DLBCL who are intolerant to first-line intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were informed about this study and voluntarily signed written informed consent
2. Patients were intolerant first-line intensive chemotherapy, including R-CHOP or R-DA-EPOCH: a) age≧70 years, or unfit or frail according to CGA; b) ECOG 0-2; c) measurable lesions
3. DLBCL with initial CR/PR according to 2016 WHO Classification of Tumor of Haematopoietic and Lymphoid Tissues
4. Life expectancy > 3 months
5. Normal blood count as defined as: absolute neutrophil count ≥1.0 × 10 9 /L independent of growth factor support, platelet count ≥ 100,000/mm 3 or ≥ 50,000/mm 3 if bone marrow (BM) involvement independent of transfusion support in either situation Normal organ functions defined as: creatinine ≤1.5 times the upper limit of normal (ULN) or estimated Glomerular Filtration Rate (Cockroft-Gault) ≥50 ml/min/1.73m 2 , aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5× the ULN; total bilirubin ≤ 1.5 × the ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN;
6. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. - Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [Beta-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.

Exclusion Criteria:

1. Contraindication to any drug in the study
2. Seropositive for or active viral infection with HBV or HCV
3. Human immunodeficiency virus (HIV) infection
4. Any grade 3 or 4 heart disease as defined by the New York Heart Association (NYHA) functional class;
5. QTc (corrected by Fridericia formula): >480ms;
6. Prior malignancies other than lymphoma in the last 5 years with exception of currently treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix
7. If female, the patient is pregnant or breast-feeding
8. Any uncontrolled active systemic infection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival | 2 years after enrollment

SECONDARY OUTCOMES:
Overall survival | From enrollment to study completion, a maximum of 4.5 years
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Overall response rate | up to 2 year, at the end of maintenance
  ORR at treatment completion or discontinuation defined as the proportion of participants with partial response (PR) or CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator and IRC(separately)
Complete response rate | up to 2 year, at the end of maintenance
  CR rate at the end of treatment by FDG-PET defined as the proportion of participants with CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator and IRC (separately)